CLINICAL TRIAL: NCT07103629
Title: Cross-sectional Study to Evaluate the Chronic Kidney Disease Prevalence Using a Creatinine Point-of-care Tool in Brazilian Adult Patients With Known CKD Risk Factors Randomly Selected
Brief Title: Bringing Knowledge About Chronic Kidney Disease in Brazil: Filling the Gap
Acronym: Filling gap
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1691R00003
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Renal Insufficiency, Chronic
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a multicenter cross-sectional study will randomly screen kidney function in adult patients with known risk factors for chronic kidney disease (CKD) within the Brazilian general population. Kidney function will be assessed using a point-of-care creatinine test at local healthcare facilities. Patients with abnormal test results will be referred for laboratory confirmation within three months and will undergo evaluation by the local nephrology team to determine the need for follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* At least one risk factor for CKD as mentioned above.

Exclusion Criteria:

* Patients with previous diagnosis of CKD
* Patients younger than 18 years old
* Patients unable to give informed consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: dult patients with at least one risk factor for Chronic Kidney Disease (CKD) listed as follows: 1) Arterial Hypertension (HTN); 2) Diabetes Mellitus (DM); 3) Cardiovascular disease (CVD); 4) Obesity (BMI ≥ 30 kg/m²); 4) Previous acute kidney injury (AKI); 5) previous history of bilateral renal lithiasis; 6) Chronic use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs); 7) Family history of genetic kidney disease. Only patients who agree to participate and sign an informed consent form will be included in the study.
Sampling Method: Probability Sample
Enrollment: 8428 (Actual)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
CKD potential prevalence | Through study completation, an avarege 1 year
  To estimate the prevalence of Chronic Kidney Disease (CKD) in Brazil through random screening using a portable device for creatinine measurement and eGFR estimation in adult patients with risk factors for the development of CKD across the five regions of the country.

SECONDARY OUTCOMES:
Regional CKD potential prevalence | Through study completation, an avarege 1 year
  To evaluate regional differences regarding CKD prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Viviane da Silva, Principal Investigator — Sociedade Brasileira de Nefrologia
Locations (1):
- Sociedade Brasileira de Nefrologia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/